CLINICAL TRIAL: NCT07172009
Title: The Effect of Chlorhexidine Mouthwash on Postprandial Glucose Response in Healthy Individuals
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Plymouth (Other)
Responsible Party: Principal Investigator, Raul Bescos, Associate Professor in Human Nutrition & Physiology, University of Plymouth
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Supportive Care
Other Study IDs: 3275
Record Dates: First submitted 2025-09-11; First posted 2025-09-15 (Actual); Last update posted 2025-09-19 (Actual); Status verified 2025-09

CONDITIONS: Glucose Metabolism Disorders (Including Diabetes Mellitus)
MeSH Terms: conditions — Glucose Metabolism Disorders

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Chlorhexidine (Experimental)
  Interventions: Other: Chlorhexidine mouthwash
- Placebo (Placebo Comparator)
  Interventions: Other: Placebo mouthwash

INTERVENTIONS:
Other: Chlorhexidine mouthwash — Rinsing the mouth with chlorhexidine mouthwash for 2 minutes before consuming 50 g of carbohydrates
  Arms: Chlorhexidine
Other: Placebo mouthwash — Rinsing the mouth with placebo mouthwash for 2 minutes before consuming 50 g of carbohydrates
  Arms: Placebo

SUMMARY:
The digestion of carbohydrates begins in the mouth through the salivary enzyme amylase which breaks food starches into maltose and disaccharides. The mouth also has a large community of microorganisms which include bacteria, fungi, viruses and protozoa that can also assist in the digestion of carbohydrates. Mouthwashes containing antibacterial compounds such as chlorhexidine are used to kill oral bacteria, but current evidence indicates that a majority of these bacteria are essential for human health.

The aim of this study is to investigate whether chlorhexidine mouthwash can also affect the digestion of carbohydrates. At least 25 individuals will be recruited. Participants will visit the laboratory in two occasions. A saliva and blood sample (fingertip to measure blood glucose) will be taken at baseline. Then, using a randomized, cross-over and double-blind design, the participants will rinse their mouth for two minutes with a placebo or chlorhexidine mouthwash. Then, participants will eat 50 g of white bread and blood glucose will be measured (fingertips) every 30 min for the following 2 hours. Another saliva sample will be collected at the end of each test.

DETAILED DESCRIPTION:
Blood glucose is measured at baseline and following food intake using a blood glucose meter (ACCU-CHEK Performa, Roche, USA). Participants are then provided with 10 mL of the assigned mouthwash according to randomisation. Mouthwashes are blinded for both researchers and participants, as they are prepared by an external individual, covered, and labelled with group numbers. This ensures that neither participants nor researchers can identify the treatment allocation.

Oral rinsing is performed for 2 minutes before participants spit out the mouthwash. The mouthwashes used include:

Chlorhexidine di-gluconate (0.2%) (Corsodyl, GlaxoSmithKline, England) Placebo (water with yellow food colouring)

Following the mouth rinse, participants consume a pre-weighed breakfast meal consisting of 40 g of Hubbard's Foodstore® strawberry jam (Sainsbury's Supermarkets Ltd., London, UK) spread over 50 g of soft white bread (Sainsbury's Supermarkets Ltd., Northern Ireland, UK).

Blood glucose measurements are taken at 15, 30, 45, 60, 90, and 120 minutes post-meal.Baseline blood glucose values are used as reference points. For analysis, only the differences between baseline and subsequent time-point measurements are considered. The mean iAUC is calculated for each mouthwash condition (chlorhexidine and placebo).

Each participant completes the protocol twice, once for each mouthwash condition, with a minimum washout period of 48 hours between sessions.

ELIGIBILITY:
Inclusion Criteria: Healthy adults (> 18 years/old)

Exclusion Criteria:

The main exclusion criteria is pregnancy, people following cancer treatment, taking immunosuppressant or antibiotics and using antibacterial mouthwash for less than 2 weeks before the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2022-06-08 (Actual); Primary Completion 2025-12-10 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Blood glucose | 2 hours

CONTACTS AND LOCATIONS:
Overall Officials: Raul Bescos Garcia, Principal Investigator — University of Plymouth
Locations (1):
- University of Plymouth, Plymouth, Devon, United Kingdom